CLINICAL TRIAL: NCT02317380
Title: Self-Affirmation and Defensiveness to Health Messages for the Self vs. a Close Other
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915034; 15-C-N034
Record Dates: First submitted 2014-12-13; First posted 2014-12-16 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09-18

CONDITIONS: Ego; Social Science; Cancer Prevention
Keywords: Self-Affirmation; Weight Loss; Self vs. Other; Cancer Risk and Prevention
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Researchers want to learn about people s beliefs and values. They also want to learn about how people respond to information about cancer risk. They have created two short studies. They have combined these studies for convenience.

Objective:

- To learn about people s beliefs and values, and about how people respond to information about cancer risk.

Eligibility:

- Adults age 40-70 who are overweight, have never had cancer, and have an opposite-sex close relationship with someone in that age group who is also overweight.

Design:

* This study will take place online or in a laboratory.
* Participants will take part in two studies. One is Values Study. The other is Cancer Risk Information.
* In Values Study, some participants will choose the most important value from a list. They will write about why that value is important to them. Others will choose the least important value from a list. They will write about why that value may be important to someone else.
* In Cancer Risk Information, participants will read a health message about a cancer risk relevant to themselves or to a close other. Some will wear special glasses that track their eye movements as they read.
* Participants will then answer questions about their beliefs about cancer risk and their intentions to lose weight.
* Both studies will take 30 minutes.

DETAILED DESCRIPTION:
Self-affirmation, a process by which individuals reflect on cherished personal values is a potent means of augmenting the effectiveness of threatening health communications. Individuals tend to be defensive against information suggesting their behavior puts them at risk for disease or negative health. Previous evidence suggests that self-affirmation may reduce defensiveness to threatening health information, increasing openness to the message and resulting in increased disease risk perceptions, disease-related worry, intentions to engage in preventive behavior, and actual behavioral change. One mechanism by which self-affirmation may be effective is by reducing self-focus and expanding self-concept. If this is the case, self-affirmation may not be effective in reducing defensiveness against information that is threatening to one s close other. We are proposing two studies to examine whether self-affirmation is equally effective at reducing defensiveness against threatening information for the self and for a close other. These studies will not only highlight conditions under which self-affirmation is effective, but also shed light on mechanisms underlying the effect.

ELIGIBILITY:
* INCLUSION CRITERIA

For Study 1

-Knowledge Networks panel members will be eligible if they are aged 40-70, overweight, and

have never been diagnosed with cancer (to ensure relevance to breast and prostate cancer risk, the topic of

the health message). Individuals will also be screened for inclusion based on whether they report having

an opposite-sex close relationship with another adult age 40-70 who is also overweight (e.g., opposite-sex

spouse, close friend, or family member).

For Study 2

-Community individuals will be subject to the same inclusion criteria.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2014-12-13; Primary Completion 2015-11-10 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Intentions to lose weight/ talk to doctor | Immediately post-experiment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Ferrer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Crocker J, Niiya Y, Mischkowski D. Why does writing about important values reduce defensiveness? Self-affirmation and the role of positive other-directed feelings. Psychol Sci. 2008 Jul;19(7):740-7. doi: 10.1111/j.1467-9280.2008.02150.x. PMID 18727791
- [Background] Epton T, Harris PR. Self-affirmation promotes health behavior change. Health Psychol. 2008 Nov;27(6):746-52. doi: 10.1037/0278-6133.27.6.746. PMID 19025270
- [Background] Godolphin W. Shared decision-making. Healthc Q. 2009;12 Spec No Patient:e186-90. doi: 10.12927/hcq.2009.20947. PMID 19667767